CLINICAL TRIAL: NCT01154452
Title: A Phase 1B/II Study of GDC-0449 (NSC 747691) in Combination With RO4929097, a Gamma-Secretase Inhibitor (GSI) in Advanced/Metastatic Sarcomas
Brief Title: Vismodegib and Gamma-Secretase/Notch Signalling Pathway Inhibitor RO4929097 in Treating Patients With Advanced or Metastatic Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01412; NCI-2011-01412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000680558; MSKCC-10049; 10-049 (Other: Memorial Sloan-Kettering Cancer Center); 8406 (Other: CTEP); N01CM62206 (NIH); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Adult Alveolar Soft Part Sarcoma; Adult Angiosarcoma; Adult Desmoplastic Small Round Cell Tumor; Adult Epithelioid Hemangioendothelioma; Adult Epithelioid Sarcoma; Adult Extraskeletal Myxoid Chondrosarcoma; Adult Extraskeletal Osteosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Liposarcoma; Adult Malignant Mesenchymoma; Adult Malignant Peripheral Nerve Sheath Tumor; Adult Rhabdomyosarcoma; Adult Synovial Sarcoma; Adult Unclassified Pleomorphic Sarcoma; Chondrosarcoma; Clear Cell Sarcoma of the Kidney; Conjunctival Kaposi Sarcoma; Dermatofibrosarcoma Protuberans; Gastrointestinal Stromal Tumor; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Osteosarcoma; Ovarian Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Adult Unclassified Pleomorphic Sarcoma of Bone; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Kaposi Sarcoma; Recurrent Osteosarcoma; Recurrent Uterine Corpus Sarcoma; Small Intestine Leiomyosarcoma; Stage III Adult Soft Tissue Sarcoma; Stage III Uterine Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Uterine Sarcoma; Unclassified Pleomorphic Sarcoma of Bone
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Hemangioendothelioma, Epithelioid; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Malignant mesenchymal tumor; Neurofibrosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Chondrosarcoma; Dermatofibrosarcoma; Gastrointestinal Stromal Tumors; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Sarcoma, Kaposi | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (gamma-secretase inhibitor RO4929097) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-21.
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (vismodegib and gamma-secretase inhibitor RO4929097) (Experimental): Patients receive vismodegib PO and gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-21.
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vismodegib

INTERVENTIONS:
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
  Arms: Arm II (vismodegib and gamma-secretase inhibitor RO4929097)

SUMMARY:
This randomized phase I/II clinical trial is studying the side effects and best dose of gamma-secretase/notch signalling pathway inhibitor RO4929097 when given together with vismodegib and to see how well they work in treating patients with advanced or metastatic sarcoma. Vismodegib may slow the growth of tumor cells. Gamma-secretase/notch signalling pathway inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vismodegib together with gamma-secretase/notch signalling pathway inhibitor RO4929097 may be an effective treatment for sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of gamma-secretase inhibitor RO4929097 (RO4929097) when given in combination with fixed-dose Hedgehog antagonist GDC-0449 (GDC-0449) which will become the recommended dose for the phase II portion of this study. (Phase Ib) II. To assess the progression-free survival (PFS) of the combination of RO4929097 with and without GDC-0449 in two arms of patients with advanced sarcoma. (Phase II)

SECONDARY OBJECTIVES:

I. To describe the tolerability and adverse event profile of daily GDC-0449 administered orally in combination with daily RO4929097 administered orally for 21 consecutive days. (Phase Ib) II. To describe the pharmacokinetics of the combination of the combination of GDC-0449 and RO4929097. (Phase Ib) III. To assess Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 overall response rates (complete and partial response [CR+PR]) for combination therapy. (Phase Ib and II) IV. To conduct pharmacodynamic studies in tissue biopsies (pre- and post-study) for explorative and hypothesis-generating studies. (Phase Ib and II) V. To assess overall survival. (Phase II) VI. To further describe the pharmacokinetics and pharmacodynamics of the combination of GDC-0449 and RO4929097 at the phase II dose at the continuous schedule. (Phase II) V. To conduct pharmacodynamic studies in tissue biopsies (pre- and post- study drug[s]) for explorative and hypothesis generating studies. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of gamma-secretase/notch signalling pathway inhibitor RO4929097 followed by a phase II study.

PHASE IB:

PART A: Patients receive vismodegib orally (PO) once daily (QD) on days 1-21.

PART B: Beginning within 7 days of finishing part A, patients receive vismodegib PO and gamma-secretase/notch signalling pathway inhibitor RO4929097 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gamma-secretase/notch signalling pathway inhibitor RO4929097 PO QD on days 1-21.

ARM II: Patients receive vismodegib PO and gamma-secretase/notch signalling pathway inhibitor RO4929097 PO QD on days 1-21.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed sarcoma
* All Patients must have measurable disease as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* There is a minimum of 1 prior therapy; however, there are no minimum systemic therapy requirements for well differentiated or de-differentiated liposarcoma, clear cell sarcoma, chondrosarcoma, alveolar soft part sarcoma and chordomas which have no effective therapies; for Phase Ib, there are no maximum limits to number of prior therapies; for Phase II, there is a maximum of 5 prior chemotherapy regimens including tyrosine kinase inhibitors (TKI); the last dose of systemic therapy (including TKI) must have been given at least 2 weeks prior to initiation of therapy; patients receiving nitrosourea (such as BCNU) or mitomycin C must have received their last dose of such therapy at least 6 weeks prior to initiation of therapy; patients receiving bevacizumab must wait at least 4 weeks; patients receiving experimental immunotherapy or antibody based therapies must wait a minimum of 4 weeks or 4 half-lives, whichever is longer; this should be discussed with the principal investigator before registration; tumor biopsies should be performed only after meeting these requirements; patients should recover to less than Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to previous therapies to be eligible
* Patients with metastatic or locally advanced (inoperable) gastrointestinal stromal tumor (GIST) must have progressed on imatinib and sunitinib or be intolerant to both drugs; the last dose of tyrosine kinase inhibitors imatinib or sunitinib should be given at least 2 weeks prior to initiation of therapy
* Patients with brain metastasis that have been treated with definitive surgery or radiation and have been clinically stable for 3 months following the procedure with no neurological signs or symptoms and no requirement for systemic glucocorticoids are eligible for study
* Patients must not have current evidence of another malignancy except non-melanoma skin cancer and superficial bladder cancer
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dl
* Platelets >= 100,000/mcL
* Total bilirubin =< upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X upper limit of normal
* Creatinine =< 1.5 or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above 1.5
* Patients treated at Memorial Sloan-Kettering Cancer Center may consent to optional tumor biopsies before and after initiation of study drug; tumor biopsies should be obtained after fulfilling requirements
* Women of child-bearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women of childbearing potential are required to have a negative pregnancy test (with a sensitivity of at least 25 mIU/mL) within 7 days and within 24 hours prior to the first dose of GDC-0449 and/or RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 3 weeks to all women of childbearing potential, at the start of each drug cycle; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449 and/or RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm that patient understands the teratogenic potential of GDC-0449 and/or RO4929097

  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months.
    * The patient is post-menopausal defined by amenorrhea for at least 1 year in a woman > 45 years old
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not receive other investigational agents within 2 weeks of enrollment in this study; patients treated with bevacizumab should be off therapy for 4 weeks; other experimental or immuno therapies should wait for 4 half-lives or 4 weeks, whichever is longer; prior exposure to Notch or Hedgehog inhibitors is not allowed; patients who have not recovered to less than CTCAE grade 2 from prior therapies are ineligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or RO4929097 used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible; patients on warfarin may be considered for enrollment after cessation of warfarin and appropriate transition to alternate anti-coagulation agents
* Preclinical studies indicate that RO4929097 is a substrate of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; the following medications with strong potential for interaction are not allowed: indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone
* Caution should be exercised when dosing GDC-0449 concurrently with medications that are substrates of cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8), CYP2C9, and CYP2C19 and have narrow therapeutic windows; caution should be exercised when dosing GDC-0449 concurrently with inhibitors of CYP3A4
* Patients must be able to swallow pills; patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* Patients with clinically active liver disease, including active viral or other hepatitis or cirrhosis, are ineligible
* Patients with uncontrolled electrolyte abnormalities including hypophosphatemia, hypocalcemia, hypomagnesemia, hyponatremia or hypokalemia or defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, a history of torsades de pointes or other significant cardiac arrhythmias that require antiarrhythmics or other medications known to prolong corrected QT interval (QTc); psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449 and/or RO4929097
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Cardiovascular: baseline QTc > 450 msec (male) or QTc > 470 msec (female)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal Gounder, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RO4929097 10mg: RO4929097: 10mg PO QD, GDC-0449: 150 mg PO QD
- RO4929097 15 mg: RO4929097: 15 mg PO QD, GDC-0449: 150 mg PO QD
- ARM 1 - RO4929097: 15 mg PO QD: ARM 1 - RO4929097: 15 mg PO QD
- ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD: ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD
Period: Phase Ib
Arm/Group | RO4929097 10mg | RO4929097 15 mg | ARM 1 - RO4929097: 15 mg PO QD | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD
Started | 6 | 4 | 0 | 0
Completed | 3 | 3 | 0 | 0
Not Completed | 3 | 1 | 0 | 0
Not completed — Not Treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0
Period: Phase II
Arm/Group | RO4929097 10mg | RO4929097 15 mg | ARM 1 - RO4929097: 15 mg PO QD | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD
Started | 0 | 0 | 35 | 33
Completed | 0 | 0 | 30 | 27
Not Completed | 0 | 0 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RO4929097 10mg | RO4929097 15 mg | ARM 1 - RO4929097: 15 mg PO QD | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD | Total
Number analyzed (Participants) | 6 | 4 | 35 | 33 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 25 | 27 | 61
  >=65 years | 0 | 1 | 10 | 6 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 15 | 15 | 34
  Male | 4 | 2 | 20 | 18 | 44
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 35 | 33 | 78

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of Gamma-secretase Inhibitor RO4929097, Defined as the Dose Level Where no More Than 1 Out of 6 Patients Experience DLT at the Highest Dose Level Below the MAD, Graded According to NCI-CTCAE Version 4.0 (Phase Ib)
Time Frame: Up to 28 days
Measure: Number; unit: mg
Groups:
- All Phase Ib Participants: All Phase Ib Participants
Arm/Group | All Phase Ib Participants
Number analyzed (Participants) | 10
mg | 15

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) of the combination of RO4929097 with and without GDC-0449 in patients with advanced sarcoma. (Phase II)
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Gamma-secretase Inhibitor RO4929097) | Arm II (Vismodegib and Gamma-secretase Inhibitor RO4929097)
Number analyzed (Participants) | 35 | 33
percentage of participants | 60 | 60

3. Secondary Outcome: Response Rate (CR + PR) as Assessed by RECIST 1.1 (Phase Ib and II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Up to 4 months
Measure: Number; unit: participants
Arm/Group | RO4929097 10mg | RO4929097 15 mg | ARM 1 - RO4929097: 15 mg PO QD | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD
Number analyzed (Participants) | 3 | 3 | 30 | 27
participants
  Stable Disease | 2 | 2 | 17 | 16
  Progression of Disease | 1 | 1 | 13 | 11

ADVERSE EVENTS:
Arm/Group | RO4929097 10mg | RO4929097 15 mg | ARM 1 - RO4929097: 15 mg PO QD | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/4 | 11/35 | 8/33
Other Adverse Events (participants affected / at risk) | 4/6 | 4/4 | 26/35 | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO4929097 10mg (N=6) | RO4929097 15 mg (N=4) | ARM 1 - RO4929097: 15 mg PO QD (N=35) | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD (N=33)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO4929097 10mg (N=6) | RO4929097 15 mg (N=4) | ARM 1 - RO4929097: 15 mg PO QD (N=35) | ARM 2: GDC-0449 150 mg PO QD and RO4929097 15 mg PO QD (N=33)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (12) | 3 (42) | 11 (56) | 8 (32)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 6 (34) | 5 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (11) | 3 (18) | 9 (21) | 4 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (13) | 1 (2) | 7 (13) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4) | 3 (26) | 14 (50) | 12 (26)
Lymphocyte count decreased (Investigations) | 2 (3) | 3 (12) | 6 (32) | 2 (5)
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 2 (3)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (6) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 3 (20) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Roche has discontinued further development of the Notch inhibitor (RO4929097) and this Phase II trial was prematurely closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less